CLINICAL TRIAL: NCT05643196
Title: A Sham-Controlled Pilot Trial of Focused Ultrasound Modulation of the Globus Pallidus Interna in Schizophrenia
Brief Title: Focused Ultrasound Modulation of the Globus Pallidus Interna in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: The New York Community Trust (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-00997
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Schizophrenia Schizoaffective
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pulsed Low-Intensity Focused Ultrasound (PLIFUS), then Sham (Experimental): Participants will receive PLIFUS sonication on the first intervention visit, then sham sonication on the second intervention visit. Visits will be separated by 1 week. Sonication at both visits will be preceded and followed by fMRI and an exit medical examination. Sonication will be delivered in a pulse pattern over 10 minutes.
  Interventions: Device: PLIFUS; Device: Sham PLIFUS; Device: MRI
- Sham, then Pulsed Low-Intensity Focused Ultrasound (PLIFUS) (Experimental): Participants will receive sham sonication on the first intervention visit, then PLIFUS sonication on the second intervention visit. Visits will be separated by 1 week. Sonication at both visits will be preceded and followed by fMRI and an exit medical examination. Sonication will be delivered in a pulse pattern over 10 minutes.
  Interventions: Device: PLIFUS; Device: Sham PLIFUS; Device: MRI

INTERVENTIONS:
Device: PLIFUS — The Sonicator-1000 system will non-invasively deliver ultrasound sonications transcranially that selectively target specific areas of the brain using a neuronavigation system and the participant's MRI brain scan. The sonication parameters follow FDA and Electrotechnical Technical Commission regulation standards for diagnostic and therapeutic ultrasound.
  Other Names: Sonicator-1000
Device: Sham PLIFUS — Sham PLIFUS treatment delivers noise and patient experience that is identical to PLIFUS with Sonicator-1000 system.
Device: MRI — A total of 5 MRIs will be performed using a Siemens 3T Prisma; one prior to the intervention visit, and one preceding and one immediately after each of the two sonication/sham visits.
  Other Names: Siemens 3T Prisma

SUMMARY:
This is a single-site, phase 2, sham-controlled random-order cross-over pilot trial of PLIFUS targeting the right GPi in individuals with schizophrenia. Twelve individuals with schizophrenia who report continuous hallucinations or delusions of mild or greater severity will receive one session of PLIFUS and one session of sham PLIFUS in random order, one week apart. If no effect of PLIFUS is detected on measures of functional connectivity or psychotic symptoms in the first four completers, the trial will be changed to 3 sessions of PLIFUS or sham administered over 5 days.

DETAILED DESCRIPTION:
The primary objectives of this study are to examine the tolerability of pulsed low-intensity focused ultrasound (PLIFUS) and its effects on brain function measured via fMRI functional connectivity and symptom response in individuals with schizophrenia. A neuronavigated single-element piezoelectric device will be utilized to noninvasively deliver transcranial PLIFUS sonication to the right globus pallidus interna, a brain region implicated in schizophrenia. The goal of this pilot study is to establish feasibility and tolerability and to determine whether the sonication procedure produces effects on the imaging biomarker and on symptoms prior to proceeding to therapeutic trials using repeated administration.

ELIGIBILITY:
Inclusion Criteria:

1. Must report current psychosis, as defined by a score of > 4 on one of the following psychosis items on the Brief Psychiatric Rating Scale (BPRS): suspiciousness, hallucinations, unusual thought content, or grandiosity continuously for at least 4 weeks.
2. Must have a diagnosis of either schizophrenia or schizoaffective disorder as established by a Structured Clinical Interview for DSM-V (SCID).
3. If taking antipsychotic medication, the dose must be unchanged for at least 4 weeks prior to randomization. If not taking antipsychotic medication, must be intending not to start medication until after completion of the study (approximately 2 weeks)-this decision must be judged to be appropriate by the research psychiatrist and by the participant's clinician.
4. If assigned female at birth and of childbearing potential, patients must

   * have a negative urine pregnancy test (all participants assigned female at birth regardless of childbearing potential will be required to submit a pregnancy test), AND;
   * not be nursing or planning a pregnancy for the duration of the study through 30 days after the last sonication visit, AND;
   * be abstinent or willing to use a reliable method of birth control from the Screening Visit and continue with the same method until termination from the study.

Exclusion Criteria:

1. Current substance abuse / dependence for substances other than nicotine and THC, (i.e. alcohol, amphetamines, barbiturates, etc.)

   * A positive urine toxicology screen (excluding THC, tricyclic antidepressants, or benzodiazepines (if prescribed).
   * Moderate or severe cannabis use disorder.
2. Diagnosis of major mood disorder or other Axis I disorder other than schizophrenia, schizoaffective disorder or schizophreniform disorder.
3. Current or recent suicidal ideation-- suicidal ideation with intent or plan (indicated by affirmative answers to items 4 or 5 of the Suicidal Ideation section of the baseline C-SSRS) in the 6 months prior to screening or subjects who represent a significant risk of suicide in the opinion of the investigator or a history of suicide attempt.
4. History of violence assessed by the Buss-Perry Aggression Questionnaire 45 and defined by violent physical contact or threat with a weapon.
5. Pregnant or nursing or positive urine pregnancy test.
6. Significant medical or neurological illness by history or physical exam, including seizure disorder, history of loss of consciousness lasting more than 30 minutes related to head trauma or intellectual developmental disorder.
7. Contraindication to MRI: Metal implants, pacemaker, or other metal in the body or piercings that cannot be removed, or claustrophobia. Individuals with tattoos will be excluded from imaging if tattoos cover more than 5% of the body surface, if a tattoo is greater than 20 cm, or if a tattoo is located on the face, neck or genitals. Individuals with a contraindication to MRI may participate in the trial but will be excluded from the elective MRI component.
8. A history or brain surgery .
9. History of syncopal episode within the past 6 months.
10. A cardiac pacemaker or intra-cardiac lines.
11. An implanted neurostimulator.
12. Implanted medication infusion device.
13. Implanted metal devices or large ferromagnetic fragments in the head or upper body (excluding dental wire), or jewelry/piercing that cannot be removed.
14. Cochlear implants.
15. Skin disease at intended stimulation sites
16. The consumption of more than four alcoholic units within 24 hours before participation or any recreational drugs within 48 hours before participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Goff, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Brooklyn, Brooklyn, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: [donald.goff@nyulangone.org]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to donald.goff@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pulsed Low-Intensity Focused Ultrasound (PLIFUS), Then Sham | Sham, Then Pulsed Low-Intensity Focused Ultrasound (PLIFUS)
Started | 5 | 5
Participants Started Treatment Period 1 (PLIFUS for Arm 1, Sharm for Arm 2) | 5 | 5
Participants Completed Treatment Period 1 (PLIFUS for Arm 1, Sharm for Arm 2) | 5 | 5
Participants Started Treatment Period 2 (Sham for Arm 1, PLIFUS for Arm 2) | 5 | 5
Participants Completed Treatment Period 2 (Sham for Arm 1, PLIFUS for Arm 2) | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pulsed Low-Intensity Focused Ultrasound (PLIFUS), Then Sham | Sham, Then Pulsed Low-Intensity Focused Ultrasound (PLIFUS) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (6.67) | 37.4 (12.9) | 38.7 (9.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 0 | 5
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 0 | 1 | 1
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Globus Pallidus Interna (GPi) Functional Connectivity During PLIFUS Intervention Visit
Description: Change in GPi functional connectivity measured via functional MRI (fMRI) captured pre-sonication and 10 minutes post-sonication during the PLIFUS intervention visit.
Time Frame: Immediately pre-sonication and 10 minutes post-sonication at Intervention Visit 1 (Day 0) and Intervention Visit 2 (Day 7)
Population: No participants were analyzed for this measure/no outcome measure data collected. The reason why this outcome did not have data collected was because there was a software issue with the scanner which made the data not analyzable. No data were collected, nor will any data be collected in relation to this outcome measure.
Groups:
- Sham: Sham PLIFUS: Sham PLIFUS treatment delivers noise and patient experience that is identical to PLIFUS with Sonicator-1000 system.
Arm/Group | PLIFUS | Sham
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Auditory Hallucinations Rating Scale (AHRS) Score From Baseline
Description: A 7-item scale developed to measure specific characteristics of auditory hallucinations (frequency, reality, loudness, number of voices, length, attentional salience, distress level). Each item is rated on a separate Likert scale. The total score, ranging from 0 to 44, indicates the overall severity of the hallucinations, with higher scores suggesting more severe symptoms.
Time Frame: Baseline, Final Study Visit (Day 14-16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIFUS | Sham
Number analyzed (Participants) | 10 | 10
score on a scale | -1.4 (2.4) | -1 (1.9)

3. Secondary Outcome: Change in Delusions Experience Sampling Assessment (DESA) Score From Baseline
Description: A 4-item scale (conviction, distress, preoccupation, disruption) used to assess moment-to-moment experience and detect more rapid changes of delusions. Participants are asked to rate the same delusional belief at the moment on a 7-point Likert scale (1 (not at all) to 7 (very much)). The total score is the sum of responses ranging from 1-28; higher scores indicate more severe symptoms.
Time Frame: Baseline, Final Study Visit (Day 14-16)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PLIFUS | Sham
Number analyzed (Participants) | 10 | 10
score on a scale | -1 (3.4) | 0.3 (2.9)

ADVERSE EVENTS:
Time Frame: AE data was collected for all events with start dates occurring any time after informed consent was obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation.
Description: Systematic Assessment for Treatment Emergent Side Effects (SAFTEE) + addendum to the SAFTEE used to assess the following side effects that have been reported in other human subject ultrasound studies: mood deterioration, scalp heating, anxiety, neck pain, and pruritis.
  Schedule: Pre/post-PLIFUS/sham at Intervention Visit 1 (Day 0); Intervention Visit 1B (Day 1-2); Pre/post-PLIFUS/sham at Intervention Visit 2 (Day 6-8); Intervention Visit 2B (Day 7-9); Final Study Visit (Day 14-16)
Arm/Group | PLIFUS | Sham
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLIFUS (N=10) | Sham (N=10)
Abnormal muscle movement (Nervous system disorders) | 0 | 1
Alcohol craving (Psychiatric disorders) | 0 | 1
Anxiety/worry (Psychiatric disorders) | 2 | 0
Appetite increase (Gastrointestinal disorders) | 0 | 1
Ataxia/impaired coordination (Nervous system disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Delusion (Psychiatric disorders) | 2 | 2
Derealization (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness/faintness (Nervous system disorders) | 1 | 1
Excitement/nervousness (Psychiatric disorders) | 1 | 0
Fatigue/weakness (General disorders) | 3 | 1
Hallucinations (Psychiatric disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 2
Insomnia (Nervous system disorders) | 0 | 2
MoCA Total Score Decrease (Nervous system disorders) | 0 | 1
Mood deterioration (Psychiatric disorders) | 0 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea/vomiting (Gastrointestinal disorders) | 0 | 2
Sedation/drowsiness (Nervous system disorders) | 0 | 2
Sensory perception abnormality (Nervous system disorders) | 0 | 1
Stomach/abdominal discomfortg (Gastrointestinal disorders) | 1 | 1
Tachycardia/palpitations (Cardiac disorders) | 1 | 0
Tinnitus/difficulty hearing (Ear and labyrinth disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT05643196/Prot_SAP_000.pdf